CLINICAL TRIAL: NCT04885348
Title: The Effectiveness of Dental Health Home Visits on Caries Prevention in Young Children - a Randomised Controlled Trial
Brief Title: The Effectiveness of Dental Health Home Visits on Caries Prevention in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Education, Malaysia (Other Government)
Responsible Party: Principal Investigator, Professor Allan Pau, Principal investigator, Ministry of Education, Malaysia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IMU R 157/2014 (FRGS)
Record Dates: First submitted 2021-05-01; First posted 2021-05-13 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Dental Caries in Children
Keywords: Dental Caries; Dental Health Home Visits; Young Children; Dental Decay
MeSH Terms: conditions — Dental Caries | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dental Home Visits and Dental Home Education Leaflets (Experimental): Two trained dental home visitors made 6-monthly Dental Home Visits (DHVs) to families in the Intervention Group. Dental Home Education Leaflets (DHELs) and oral health messages were delivered through a personalized approach that avoids direct persuasion.
  Interventions: Behavioral: Intervention Group (Dental Home Visits + Dental Home Education Leaflets); Behavioral: Control Group (Dental Home Education Leaflets)
- Dental Home Education Leaflets (Active Comparator): Only Dental Home Education Leaflets were provided every six months for 2 years.
  Interventions: Behavioral: Control Group (Dental Home Education Leaflets)

INTERVENTIONS:
Behavioral: Intervention Group (Dental Home Visits + Dental Home Education Leaflets) — No drugs were given in the Intervention. The intervention group received Dental Home Visits consisted of 6 monthly home visits by oral health therapists/dental home visitors where they deliver dental care advice to the parents for durations of approximately 30 minutes until follow-up at two years. Dental Home Education Leaflets (DHELs) and oral health messages were delivered through a personalized approach that avoids direct persuasion. These messages included information on daily tooth brushing with fluoride toothpaste, controlling dietary sugar intake, and the need for regular dental check-ups. The families were also be provided with information about local dental services available in their vicinity and how to access these services.
  Arms: Dental Home Visits and Dental Home Education Leaflets
Behavioral: Control Group (Dental Home Education Leaflets) — Only Dental Home Education Leaflets were provided every six months for 2 years.

SUMMARY:
Tooth decay affects 75% of Malaysian preschool children, most of which remain untreated. Untreated decay can cause pain, and impair nutritional status and physical growth. In 2012, nearly 4,000 children in Malaysia were referred for hospital paediatric dental services because of early childhood caries. The realistic management of these children would have been treatment under general anaesthesia or sedation, at considerable cost to the state, and distress to the children and families. The amount of dental disease in young children who have been referred to the hospital children's dentistry service for severe caries is disturbing, particularly given the fact that each district has a dental clinic and that the water is very likely to be fluoridated. It is unlikely that there will ever be enough dental clinics and dental practitioners to manage the amount of disease. Clearly, existing health services need to be supplemented with a population-based approach to promote child oral health. The investigators, therefore, propose a community trial study to investigate the effectiveness of a dental health visiting service for caries control in young children. It is likely that such a home-based intervention is influenced by the family dynamics in which the child lives. The investigators further propose to assess the cost-effectiveness of dental home visits (DHVs). Health economic evaluation can be used to assess health services to ensure there is cost-efficient resource allocation. Economic evaluation is defined as the comparative analysis of alternative courses of action in terms of both their costs and consequences. A health intervention is considered cost-effective when it produces acceptable costs and health benefits. Economic data are now recognized as important due to the fact that dental disease is very common and expensive for the health care system.

This study was conducted in collaboration with the National Oral Health of Pre-school Survey (NOHPS), in which a sub-sample will be followed up for two years. The NOHPS is a national survey of the oral health of 5-year-olds that takes place every 10 years.

This is a randomized controlled trial to assess the cost-effectiveness of home-based DHVs with families of children at high risk of caries in caries prevention compared to children receiving oral health information in the form of an education leaflet (ELs) alone. A collaborative project with the Oral Health Division (OHD) at the Ministry of Health is proposed. The OHD will provide access to a sub-sample from the National Oral Health Preschool Survey (NOHPS), with clinical dental health data.

ELIGIBILITY:
Inclusion Criteria:

* All the children age of 5 or 6-year-old with parents' consents to participate from these kindergartens will be included as the subjects of this study

Exclusion Criteria:

-

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 329 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Number of children developing new caries in deciduous molars. | 2 years
  The number of children developing caries in deciduous molars over the two years follow up.
Number of in deciduous molars developing new caries. | 2 years
  New caries detected in deciduous molars at the cavitation stage.

REFERENCES:
- [Background] Sheiham A. Dental caries affects body weight, growth and quality of life in pre-school children. Br Dent J. 2006 Nov 25;201(10):625-6. doi: 10.1038/sj.bdj.4814259. PMID 17128231
- [Background] M E Drummond, M J Sculpher, G W Torrance GW, et al. Oxford University Press, 2005. ISBN 0-19-852945-7
- [Background] Masood M, Yusof N, Hassan MI, Jaafar N. Assessment of dental caries predictors in 6-year-old school children - results from 5-year retrospective cohort study. BMC Public Health. 2012 Nov 16;12:989. doi: 10.1186/1471-2458-12-989. PMID 23158416
- [Background] Seow WK. Biological mechanisms of early childhood caries. Community Dent Oral Epidemiol. 1998;26(1 Suppl):8-27. doi: 10.1111/j.1600-0528.1998.tb02090.x. PMID 9671196